CLINICAL TRIAL: NCT00953017
Title: A Randomized, Blinded Trial Comparing Miralax With Amitiza Pretreatment Versus Miralax With Dulcolax Pretreatment Versus Miralax Alone Without Pretreatment Versus Golytely for Bowel Cleansing Prior to Colonoscopy
Brief Title: A Trial Comparing Split-Dose Miralax With Amitiza Pretreatment Versus Dulcolax Pretreatment Versus Golytely for Bowel Cleansing Prior to Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joel Z. Stengel, Gastroenterology Fellow, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C.2009.209
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Results first posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Colonoscopy
Keywords: Efficacy of bowel cleansing; Patient tolerability; Amitiza; Dulcolax; Miralax; Colonoscopy preparation; Bowel preparation; Screening colonoscopy
MeSH Terms: interventions — polyethylene glycol 3350; Lubiprostone; Bisacodyl; Golytely; Polyethylene Glycols

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Miralax plus Amitiza (Active Comparator): 106 patients randomized to Miralax plus Amitiza will take one 24mcg gelcap of Amitiza at noon the day prior to their colonoscopy. On the day prior to the colonoscopy, the patients will mix 255gm of Miralax with 64 oz. of Gatorade and drink 32 oz. of the solution at 4 p.m. The remaining 32 oz. of the solution will be completed the morning of the procedure, approximately 4-6 hours prior to the scheduled start time of the colonoscopy.
  Interventions: Drug: Amitiza (Lubiprostone)
- Miralax plus Dulcolax (Active Comparator): 107 patients randomized to Miralax plus Dulcolax will take two 5mg tablets of Dulcolax at noon the day prior to their colonoscopy. On the day prior to the colonoscopy, the patients will mix 255gm of Miralax with 64 oz. of Gatorade and drink 32 oz. of the solution at 4 p.m. The remaining 32 oz. of the solution will be completed the morning of the procedure, approximately 4-6 hours prior to the scheduled start time of the colonoscopy.
  Interventions: Drug: Dulcolax (Bisacodyl)
- Miralax (Active Comparator): 106 patients will mix 255gm of Miralax with 64 oz. of Gatorade and drink 32 oz. of the solution at 4 p.m. The remaining 32 oz. of the solution will be completed the morning of the procedure, approximately 4-6 hours prior to the scheduled start time of the colonoscopy.
  Interventions: Drug: Miralax (PEG 3350)
- Golytely (polyethylene glycol) (Active Comparator): 106 patients will take 1 gallon of golytley (Polyethylene glycol) and drink 1/2 of the solution at 4 p.m. The remaining 1/2 of the solution will be completed the morning of the procedure, approximately 4-6 hours prior to the scheduled start time of the colonoscopy
  Interventions: Drug: Golytely (polyethylene glycol)

INTERVENTIONS:
Drug: Miralax (PEG 3350) — Miralax 255gm bottle
  Arms: Miralax
Drug: Amitiza (Lubiprostone) — Amitiza 24mcg gelcap
  Arms: Miralax plus Amitiza
Drug: Dulcolax (Bisacodyl) — Bisacodyl 5mg tab x2
  Arms: Miralax plus Dulcolax
Drug: Golytely (polyethylene glycol) — Golytely 1 gallon
  Arms: Golytely (polyethylene glycol)

SUMMARY:
Miralax (PEG 3350) has been shown to be a safe and uncomplicated bowel preparation prior to colonoscopy in pediatric populations. This study seeks to confirm the efficacy of this bowel cleansing regimen in adults and to determine the benefit of adding a pretreatment medication to this bowel preparation. The tolerability of Miralax will hopefully improve patient satisfaction with colonoscopy and decrease their reluctance to be screened because of the uncomfortable taste and side effects of bowel preparation regimens.

ELIGIBILITY:
Inclusion Criteria:

* adult patients referred to our clinic for average or increased risk screening for colorectal cancer

Exclusion Criteria:

* elevated serum creatinine (Men >1.4mg/dL, Women >1.3mg/dL)
* previous diagnosis of congestive heart failure
* history of bowel obstruction
* history of solid organ transplant
* current pregnancy
* lactating mother
* participants allergic to either polyethylene glycol (Miralax), lubiprostone (Amitiza), or bisacodyl (Dulcolax)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

REFERENCES:
- [Derived] Hjelkrem M, Stengel J, Liu M, Jones DP, Harrison SA. MiraLAX is not as effective as GoLytely in bowel cleansing before screening colonoscopies. Clin Gastroenterol Hepatol. 2011 Apr;9(4):326-332.e1. doi: 10.1016/j.cgh.2010.11.007. Epub 2010 Nov 27. PMID 21115134

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All pateints were recruited and enrolled at Brooke Army Medical Center in San Antonio, TX from July 1, 2009 to July 1, 2010.
Pre-assignment Details: NO significant events occured prior to study participant enrollment.
Period: Overall Study
Arm/Group | Miralax Plus Amitiza | Miralax Plus Dulcolax | Miralax | Golytely (Polyethylene Glycol)
Started | 106 | 107 | 106 | 106
Completed | 101 | 101 | 100 | 101
Not Completed | 5 | 6 | 6 | 5
Not completed — DId not show up for colonoscopy | 4 | 4 | 5 | 4
Not completed — Incomplete data | 1 | 1 | 0 | 0
Not completed — Procedure incomplete due to pain/looping | 0 | 1 | 0 | 1
Not completed — Brown stool prior to procedure | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Miralax Plus Amitiza | Miralax Plus Dulcolax | Miralax | Golytely (Polyethylene Glycol) | Total
Number analyzed (Participants) | 106 | 107 | 106 | 106 | 425
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 104 | 107 | 106 | 104 | 421
  >=65 years | 2 | 0 | 0 | 2 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 55.4 (5.7) | 53.8 (5.4) | 54.1 (5.3) | 54.2 (6.7) | 54 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 48 | 54 | 49 | 206
  Male | 51 | 59 | 52 | 57 | 219
Region of Enrollment [Number; unit: participants]
  United States | 106 | 107 | 106 | 106 | 425

OUTCOME MEASURES:

1. Primary Outcome: The Cleanliness of the Prep as Measured by the Ottawa Scale
Description: Bowel cleansing was evaluated with the Ottawa bowel preparation scale by each endoscopist during the endoscopy. Neither the endoscopist nor the endoscopy nurse was aware of the bowel preparation used prior to the colonoscopy. The Ottawa bowel preparation scale is a validated tool and was used in this study to provide a reliable quality assessment of the bowel preparation used for colonoscopy. This validated scale rates each section of the colon, the right, the mid, and the rectosigmoid colon, on a 5-point scale (0-4), as well as a global 3-point rating for overall colonic fluid (0-2). The total score ranges from 0 to 14. An excellent preparation with little fluid would score 0-3, a good preparation 4-6, while scores higher than 7 would indicate progressively worsening bowel preparations. A completely unprepared colon would score 11-14, depending on the amount of colonic fluid.
Time Frame: measured at the time of colonoscopy
Measure: Mean (Full Range); unit: Ottawa Scale
Arm/Group | Miralax Plus Amitiza | Miralax Plus Dulcolax | Miralax | Golytely (Polyethylene Glycol)
Number analyzed (Participants) | 101 | 101 | 100 | 101
Ottawa Scale | 6.3 [4 to 12] | 6.8 [4 to 13] | 6.9 [4 to 13] | 5.1 [3 to 10]

2. Secondary Outcome: Patient Satisfaction With the Prep Measured by 5 Point Likert Scale
Description: patient satisfaction based on a Likert Scale from 0-5 (5 being completely satisfied and 0 being not satisfied)
Time Frame: measured at check in to colonoscopy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Miralax Plus Amitiza | Miralax Plus Dulcolax | Miralax | Golytely (Polyethylene Glycol)
Number analyzed (Participants) | 101 | 101 | 100 | 101
units on a scale | 3.8 (1.1) | 4.1 (0.8) | 4.0 (1.0) | 3.2 (1.0)

3. Secondary Outcome: Procedure Time
Description: total colonoscopy procedure time
Time Frame: measured at the time of colonoscopy
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Miralax Plus Amitiza | Miralax Plus Dulcolax | Miralax | Golytely (Polyethylene Glycol)
Number analyzed (Participants) | 101 | 101 | 100 | 101
minutes | 21.3 (10.2) | 19.3 (8.1) | 20 (9) | 18.3 (7.2)

4. Secondary Outcome: Polyps Detected
Description: Number of polyps
Time Frame: measured at the time of colonoscopy
Measure: Number; unit: polyps
Arm/Group | Miralax Plus Amitiza | Miralax Plus Dulcolax | Miralax | Golytely (Polyethylene Glycol)
Number analyzed (Participants) | 101 | 101 | 100 | 101
polyps | 128 | 92 | 90 | 101

ADVERSE EVENTS:
Time Frame: 1 year
Description: Questionnaire was used to identify all 'Other (Not Including Serious) Adverse Events'
Arm/Group | Miralax Plus Amitiza | Miralax Plus Dulcolax | Miralax | Golytely (Polyethylene Glycol)
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/101 | 0/100 | 0/101
Other Adverse Events (participants affected / at risk) | 6/101 | 4/101 | 6/100 | 7/101
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Miralax Plus Amitiza (N=101) | Miralax Plus Dulcolax (N=101) | Miralax (N=100) | Golytely (Polyethylene Glycol) (N=101)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 6 (6) | 4 (4) — questionnaire used to identify any patient complaints of nausea
Abdominal Cramping (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2) | 4 (4) — questionnaire used to identify any patient complaints of abdominal cramping
Abdominal Bloating (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) — questionnaire used to identify any patient complaints of abdominal bloating

LIMITATIONS AND CAVEATS:
Indication for colonoscopy was restricted to colorectal cancer screening. Patients admitted to the hospital were not included. Polyp detection rates could have been influenced by unequal randomization of high-risk and low-risk patients for adenomas.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes